CLINICAL TRIAL: NCT06785857
Title: An Intervention Effect Study of a Mobile Medical Supportive Care Program for Family Caregivers With Dementia Combined With Diabetes: a Randomized Controlled Trial
Brief Title: A Study of Mobile Medical Supportive Care Program for Family Caregivers With Dementia Combined With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuanjiao Yan (Other)
Responsible Party: Sponsor-Investigator, Yuanjiao Yan, Sponsor-Investigator, Fujian Provincial Hospital
Organization: Fujian Provincial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: K2021-05-024
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Diabetes; Senile Dementia, Alzheimer Type
Keywords: Dementia; Diabetes; Family caregivers; Mobile healthcare; Supportive care programs; A randomized controlled trial
MeSH Terms: conditions — Diabetes Mellitus; Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The intervention group received an mHealth supportive care program, the control group received an offline supportive care program, and all caregivers received health education related to diabetes and dementia. The intervention was conducted concurrently in the experimental and control groups, and both groups were followed up in the home once a month for 12 weeks, with each caregiver receiving three 1-hour visits from the researcher.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- an offline supportive care program (Active Comparator): This was done routinely in accordance with the requirements of public health services for chronic diseases in the community elderly. In addition, health education on diabetes mellitus and dementia was provided to the caregivers during their monthly home visits.
  ① the content of diabetes health education: the researcher gave the caregivers education and training on the care of diabetes patients: the main points of care in diet, sleep, exercise, etc.
  ② The content of dementia health education: the researcher gave the caregivers education and training related to the care of dementia patients: instructing the caregivers in the basic life care skills of patients' diet, sleep, exercise, etc.
  Interventions: Other: Offline supportive care
- mHealth Supportive Care Program (Experimental): On the basis of the monthly home visits in the control group, "Xiamen iHealth" was used as a medium to add a weekly mHealth supportive care intervention program, with one supportive care item every two weeks for 12 weeks, for a total of 12 online interventions, as well as to provide online consultation and appointment services for caregivers at any time.
  Interventions: Other: mHealth Supportive Care Program

INTERVENTIONS:
Other: mHealth Supportive Care Program — On the basis of monthly home visits in the control group, a weekly mHealth supportive care intervention program was added through the medium of Xiamen iHealth, with one supportive care item every two weeks for 12 weeks, for a total of 12 online interventions, as well as the provision of online consulting and booking services for caregivers at any time.
  Arms: mHealth Supportive Care Program
Other: Offline supportive care — This was done routinely in accordance with the requirements of public health services for chronic diseases in the community elderly. In addition, health education on diabetes mellitus and dementia was provided to the caregivers during their monthly home visits.
  ① the content of diabetes health education: the researcher gave the caregivers education and training on the care of diabetes patients: the main points of care in diet, sleep, exercise, etc.
  ② The content of dementia health education: the researcher gave the caregivers education and training related to the care of dementia patients: instructing the caregivers in the basic life care skills of patients' diet, sleep, exercise, etc.
  Arms: an offline supportive care program

SUMMARY:
The purpose of this project is to evaluate the effectiveness of the clinical application of a mHealth supportive care program for family caregivers with dementia combined with diabetes based on the supportive care framework. The results of the study will provide family caregivers with more economical and efficient care guidance, thereby improving the quality of care and quality of life for people with dementia and diabetes in general.

ELIGIBILITY:
Inclusion Criteria:

Caregivers:

* caregivers and patients have legal kinship (such as spouses, children or siblings) and other non-costly caregivers such as babysitters, bellhops, etc.;
* caregiving work ≥ 8 hours / day, care for the patient ≥ 5 days a week, the care time ≥ 1 month;
* conscious adults with a certain degree of reading and comprehension;
* at least have a smart phone (with Internet access) and will be able to use it proficiently;
* informed consent and voluntary participation in the study. Informed consent and voluntary participation in the study.

Targets:

* meet the diagnostic criteria of Alzheimer's disease;
* meet the diagnostic criteria of type 2 diabetes mellitus;
* age ≥ 60 years old, permanent residents of the district.

Exclusion Criteria:

Caregivers:

* severe physical or mental illness;
* people with drug or alcohol dependence;
* caregivers who are participating in a similar intervention study.

Caregivers:

* patients with severe physical illnesses, major illnesses, or terminal illnesses;
* patients with drug or alcohol dependence.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Community Health Center, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Research data and research-related materials will be available in a repository or online. After completion of the study, relevant data will be provided in the form of a URL or DOI.
Supporting Information: SAP, Analytic Code
Time Frame: After completion of the study,relevant data will be provided in the form of a URL or DOI.
Access Criteria: Researchers whose proposed use of the data has been approved.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolls family caregivers of elderly patients with both dementia and type 2 diabetes. The patients themselves are not active participants in the study. Their diagnostic criteria (e.g., dementia, diabetes, age ≥60) are solely used to define eligibility for their caregivers. All study procedures (interventions, data collection, and outcome measures) are directed at caregivers only. Patients do not receive interventions or undergo study assessments.
Pre-assignment Details: The total enrollment number (N=60) refers to individual caregivers (not patient-caregiver dyads). Collected only for caregivers (e.g., demographics, Caregiver Burden Inventory [CBI], Social Support Rating Scale [SSRS]). Patient data (e.g., diagnosis confirmation) were used only for screening. All outcomes (e.g., caregiver burden, knowledge, social support) are caregiver-centered. No patient health outcomes are measured.
Groups:
- mHealth Supportive Care Program: Caregivers were randomly assigned to the intervention group. On the basis of the monthly home visits in the control group, "Xiamen iHealth" was used as a medium to add a weekly mHealth supportive care intervention program, with one supportive care item every two weeks for 12 weeks, for a total of 12 online interventions, as well as to provide online consultation and appointment services for caregivers at any time.
  mHealth Supportive Care Program: On the basis of monthly home visits in the control group, a weekly mHealth supportive care intervention program was added through the medium of Xiamen iHealth, with one supportive care item every two weeks for 12 weeks, for a total of 12 online interventions, as well as the provision of online consulting and booking services for caregivers at any time.
- an Offline Supportive Care Program: Caregivers were randomly assigned to the control group. This was done routinely in accordance with the requirements of public health services for chronic diseases in the community elderly. In addition, health education on diabetes mellitus and dementia was provided to the caregivers during their monthly home visits.
  ① the content of diabetes health education: the researcher gave the caregivers education and training on the care of diabetes patients: the main points of care in diet, sleep, exercise, etc.
  ② The content of dementia health education: the researcher gave the caregivers education and training related to the care of dementia patients: instructing the caregivers in the basic life care skills of patients' diet, sleep, exercise, etc.
  Offline supportive care: This was done routinely in accordance with the requirements of public health services for chronic diseases in the community elderly. In addition, health education on diabetes mellitus and dementia was provided to the caregivers during their monthly home visits.
  ① the content of diabetes health education: the researcher gave the caregivers education and training on the care of diabetes patients: the main points of care in diet, sleep, exercise, etc.
  ② The content of dementia health education: the researcher gave the caregivers education and training related to the care of dementia patients: instructing the caregivers in the basic life care skills of patients' diet, sleep, exercise, etc.
Period: Overall Study
Arm/Group | mHealth Supportive Care Program | an Offline Supportive Care Program
Started | 30 | 30
Completed | 28 | 27
Not Completed | 2 | 3
Not completed — Death of the Care recipient (Patients with Dementia and TDM2) | 2 | 3

BASELINE CHARACTERISTICS:
Population: Family caregivers was randomly allocated in a strict 1:1 ratio at baseline, with 30 carers in each of the intervention and control groups (60 cases in total). During the course of the intervention, 2 carers in the intervention group withdrew from the study due to the death of the care recipient (patient) and 3 in the control group withdrew for the same reason. Therefore, the final number of participants who completed the analysis was 28 in the intervention group and 27 in the control group.
Groups:
- an Offline Supportive Care Program: This was done routinely in accordance with the requirements of public health services for chronic diseases in the community elderly. In addition, health education on diabetes mellitus and dementia was provided to the caregivers during their monthly home visits.
  ① the content of diabetes health education: the researcher gave the caregivers education and training on the care of diabetes patients: the main points of care in diet, sleep, exercise, etc.
  ② The content of dementia health education: the researcher gave the caregivers education and training related to the care of dementia patients: instructing the caregivers in the basic life care skills of patients' diet, sleep, exercise, etc.
  Offline supportive care: This was done routinely in accordance with the requirements of public health services for chronic diseases in the community elderly. In addition, health education on diabetes mellitus and dementia was provided to the caregivers during their monthly home visits.
  ① the content of diabetes health education: the researcher gave the caregivers education and training on the care of diabetes patients: the main points of care in diet, sleep, exercise, etc.
  ② The content of dementia health education: the researcher gave the caregivers education and training related to the care of dementia patients: instructing the caregivers in the basic life care skills of patients' diet, sleep, exercise, etc.
- Total: Total of all reporting groups
Arm/Group | an Offline Supportive Care Program | mHealth Supportive Care Program | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Customized [Count of Participants; unit: Participants] — Population: Withdrawal due to death of the care recipient.
  Participants
    Age (years): <60 | 11 | 16 | 27
    Age (years): ≥ 60 | 16 | 12 | 28
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Withdrawal due to death of the care recipient.
  Participants
    Female | 15 | 15 | 30
    Male | 12 | 13 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Caregiver Burden Inventory (CBI) [Median (Inter-Quartile Range); unit: units on a scale] — The Caregiver Burden Inventory (CBI) was used to evaluate the burden experienced by the FCGs of individuals with dementia and diabetes. Each item is scored using a Likert 5-point scale ranging from strongly agree (4 points) to strongly disagree (0 points). The total score of the scale ranges from 0-96, with higher scores indicating a heavier caregiver burden. Scores ≥24 suggest the need for therapeutic intervention, whereas scores ≥36 indicate a risk of severe burden. Population: Withdrawal due to death of the care recipient.
  units on a scale | 56.00 [53.00 to 60.00] | 57.00 [54.00 to 60.75] | 57.00 [53.00 to 60.00]
The Social Support Scale (SSRS) [Mean (Standard Deviation); unit: units on a scale] — The social support rating scale (SSRS) is a 10-item rating scale that evaluates each person's psychological support an individual receives in social life and their utilization of such support. The total score ranges from 12 to 48. Higher scores indicate higher levels of social support. Generally, scores below 20 indicate low social support, 20-30 indicate moderate social support, and 30-40 indicate satisfactory social support. Population: Withdrawal due to death of the care recipient.
  units on a scale | 24.11 (2.76) | 24.71 (1.88) | 24.42 (5.54)
The Dementia Caring Knowledge Scale (DCKS) [Median (Inter-Quartile Range); unit: units on a scale] — The dementia caring knowledge scale (DCKS) was used to assess the FCGs extent of knowledge about dementia caring. This questionnaire, based on Maslow's hierarchy of needs, covers personal hygiene, diet, excretion, sleep, disease and rehabilitation, medication, environmental and travel safety, social relationships and family ties, self-esteem, and self-actualization. The DCKS scores range from 0-22, with higher scores reflecting a higher level of dementia care knowledge. Population: Withdrawal due to death of the care recipient.
  units on a scale | 12.00 [10.00 to 16.00] | 11.00 [10.00 to 12.75] | 11.00 [10.00 to 16.00]

OUTCOME MEASURES:

1. Primary Outcome: Caregiver Burden Inventory- Baseline (Month 0)
Description: The scale used in this study was obtained by Rui Zhang based on the Chinese version of the CBI by Taiwanese scholar Guiru Zhou, who modified the questionnaire according to the linguistic characteristics of mainland China.The CBI was initially used to measure the evaluation of the burden on caregivers of patients with dementia, which includes multiple dimensions such as physical burden, emotional burden, social burden, time-dependent burden, and developmentally limited burden, and the scoring of each entry was based on a Likert 5-point scale ranging from strongly agree (4) to strongly disagree (0). Likert 5-point scale from strongly agree (4 points) to strongly disagree (0 points). Total scale scores ranged from 0 to 96; higher scores indicated greater caregiver burden. When the score is ≥ 24, consideration should be given to receiving therapeutic interventions; when the score is greater than or equal to 36, it suggests the risk of severe burden.
Time Frame: Baseline (pre-intervention)
Population: Withdrawal due to the death of the care recipient.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | an Offline Supportive Care Program | mHealth Supportive Care Program
Number analyzed (Participants) | 27 | 28
score on a scale | 56 [53 to 60] | 57 [54 to 60.75]

2. Secondary Outcome: Social Support Rating Scale - Post-intervention (Month 3)
Description: The Social Support Scale was developed by Xiao Shuiyuan, a Chinese scholar, based on China's national conditions, and contains a total of 10 scores. This scale aims to detect the degree of psychological support received by the individual in the social life, and the utilization of support. The total score ranges from 12 to 48. Higher scores indicate higher levels of social support. Generally, scores below 20 indicate low social support, 20-30 indicate moderate social support, and 30-40 indicate satisfactory social support. The re-test reliability of the scale is 0.92, and the consistency of the items is between 0.89 and 0.94; the Cronbach's alpha coefficient is 0.89.
Time Frame: Post-intervention (Month 3)
Population: Withdrawal due to the death of the care recipient.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | an Offline Supportive Care Program | mHealth Supportive Care Program
Number analyzed (Participants) | 27 | 28
score on a scale | 31 [28 to 32] | 32 [30 to 34]

3. Secondary Outcome: Dementia Caring Knowledge Scale - Post-intervention (Month 3)
Description: The Dementia Caregiver Knowledge Assessment Scale (DKAS) is based on Maslow's Hierarchy of Needs as a theoretical framework, with "yes", "no", or "don't know" answers for each item. Personal hygiene, diet, excretion, sleep, disease and rehabilitation, medication, safety of the environment and travel, social intimacy, self-esteem, self-realization, etc.; quantitative scoring method, 1 point for a correct answer, 0 points for an incorrect answer or "don't know"; the total score of the scale is 22 points, and the higher the score, the higher the knowledge of dementia caregivers about dementia care. The total score of the scale was 22 points, and the higher the score, the higher the caregiver's knowledge of dementia care; the Cronbach's alpha coefficient of the total scale was 0.626, and the content validity of the scale ranged from 0.86 to 1, with an average CVI of 0.95.
Time Frame: Post-intervention (Month 3)
Population: Withdrawal due to the death of the care recipient.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | an Offline Supportive Care Program | mHealth Supportive Care Program
Number analyzed (Participants) | 27 | 28
score on a scale | 16 [15 to 18] | 19 [18 to 19]

4. Primary Outcome: Caregiver Burden Inventory - Post-intervention (Month 3)
Description: as for outcome 1
Time Frame: Post-intervention (Month 3)
Population: Withdrawal due to the death of the care recipient.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | an Offline Supportive Care Program | mHealth Supportive Care Program
Number analyzed (Participants) | 27 | 28
score on a scale | 52 [49 to 55] | 48 [46 to 50.75]

5. Secondary Outcome: Social Support Rating Scale - Baseline (Month 0)
Description: as for outcome 2
Time Frame: Baseline (Pre-intervention)
Population: Withdrawal due to the death of the care recipient.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | an Offline Supportive Care Program | mHealth Supportive Care Program
Number analyzed (Participants) | 27 | 28
score on a scale | 24.11 (2.76) | 24.71 (1.88)

6. Secondary Outcome: Dementia Caring Knowledge Scale-Baseline (Month 0)
Description: as for outcome 3
Time Frame: Baseline (Pre-intervention)
Population: Withdrawal due to the death of the care recipient.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | an Offline Supportive Care Program | mHealth Supportive Care Program
Number analyzed (Participants) | 27 | 28
score on a scale | 12.3 (3.45) | 11.32 (2.13)

ADVERSE EVENTS:
Time Frame: 3months
Description: This study did not actively monitor or assess Serious or Other Adverse Events for caregivers, as the supportive care interventions were considered minimal risk. The participant withdrawals (Offline:3; mHealth:2) reported in All-Cause Mortality were due to the death of their care recipients (patients), not due to any adverse events or deaths among the caregivers themselves. No caregivers died or experienced reported adverse events.
Arm/Group | an Offline Supportive Care Program | mHealth Supportive Care Program
All-Cause Mortality (participants affected / at risk) | 3/30 | 2/30
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT06785857/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT06785857/ICF_001.pdf